CLINICAL TRIAL: NCT01883908
Title: A Pilot Randomized Controlled Trial to Evaluate the Efficacy and Explore the Mechanism of Acupuncture in Reducing the Severity of Chemoradiation-induced Mucositis in Patients With Oropharyngeal Cancer.
Brief Title: Acupuncture in Reducing the Severity of Chemoradiation-induced Mucositis in Patients With Oropharyngeal Cancer
Acronym: GCC1229
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The project is terminated due to that fact that the PI has moved to another institution and there are no resources to keep the study open in either institution.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00053319; GCC1229 (Other: University of Maryland Greenebaum Cancer Center)
Record Dates: First submitted 2013-03-13; First posted 2013-06-21 (Estimated); Results first posted 2015-10-07 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Mucositis; Oropharyngeal Cancer
Keywords: Acupuncture therapy; Mucositis; oropharyngeal cancer
MeSH Terms: conditions — Mucositis; Oropharyngeal Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture with Seirin® needles (Experimental): Participants will be randomized to receive acupuncture treatment plus usual medical care once a week for 8 weeks coinciding with their chemoradiation treatments. The length of the study will be 16 weeks: 8 weeks of treatment and two follow up visits at 4 weeks and 8 weeks after radiation (weeks 12 and 16).
  Interventions: Device: Acupuncture with Seirin® needles; Other: Usual medical care
- Usual medical care (Active Comparator): Participants will be randomized to receive usual medical care for 8 weeks coinciding with their chemoradiation treatments. Patients will receive usual medical care such as viscous Lidocaine for relief of pain.
  Interventions: Other: Usual medical care

INTERVENTIONS:
Device: Acupuncture with Seirin® needles — Participants will be randomized to receive either usual medical care or acupuncture treatment plus usual medical care once a week for 8 weeks coinciding with their chemoradiation treatments. The length of the study will be 16 weeks: 8 weeks of treatment and two follow up visits at 4 weeks and 8 weeks after radiation (weeks 12 and 16).
  Arms: Acupuncture with Seirin® needles
Other: Usual medical care — usual medical care such as viscous Lidocaine for relief of pain

SUMMARY:
Patients are asked to be in this study if have oropharyngeal cancer and will be treated with chemotherapy and radiation.

This research is being done to find out if acupuncture can reduce the mouth inflammation and pain caused by chemotherapy and radiation. Chemoradiation may cause mouth inflammation and pain.

Acupuncture is a medical technique of inserting very thin needles into the "energy points" on the body with the aim to restore health and well-being. It has been used widely to treat pain, such as lower back pain and joint pain. In this study we will assess the potential usefulness of acupuncture to decrease the severity of mucositis and mucositis-related mouth and throat pain in patients receiving chemoradiation for oropharyngeal cancer.

Mouth cancer patients receiving chemoradiation who have not had acupuncture within the last one month and who do not have a history of head and neck cancer may join this pilot study.

DETAILED DESCRIPTION:
This is a single-center, randomized controlled pilot clinical trial (n=20) assessing the efficacy, feasibility and safety of acupuncture in reducing the severity of chemoradiation-induced oral mucositis (CRIOM) in patients with oropharyngeal cancer. Participants will be randomized to receive either usual medical care or acupuncture treatment plus usual medical care once a week for 8 weeks coinciding with their chemoradiation treatments. The length of the study will be 16 weeks: 8 weeks of treatment and two follow up visits at 4 weeks and 8 weeks after radiation (weeks 12 and 16). All subjects will receive usual medical care in addition to the study intervention. The Oral Mucositis Daily Questionnaire for Head and Neck Cancer patients (OMDQ) will be used to assess patients' self-reported chemoradiation-induced mucositis severity at baseline (before 1st acupuncture session), and daily throughout the course of radiation, as well as at the 12 and 16 week follow up visits. At baseline, weekly during radiation therapy, and at the 12 and 16 week follow up appointments, patients will complete the Functional Assessment of Cancer Therapy (FACT-G), Esophagus Cancer subscale (ESC) QOL, and the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue subscale questionnaires. Oral mucositis will also be assessed objectively by a trained member of the research team using both the Oral Mucositis Assessment Scale (OMAS) and the National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE) v3.0 measurement scale once a week for the first two weeks of chemoradiation treatment, then twice a week during weeks three through seven, and additionally once during week 8 and once at the 12 and 16 week follow up visits. Twice weekly measurements correspond to peak severity of mucositis during weeks three to seven, based on previous reports in the literature. Patients will be given a weekly diary to record oral analgesic intake. Lastly, 8 milliliters of blood and a saliva sample will be taken from the subjects at baseline (before 1st acupuncture session), weekly through radiation treatment, and at the week 12 and 16 follow up visits to measure changes in proinflammatory cytokines concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of oropharyngeal cancer.
* The patient plans on undergoing external beam radiation with concomitant chemotherapy.
* Eastern Cooperative Group in Oncology (ECOG) performance status 0-3.
* Men and women who are ≥ 18 years old
* The patient is aware of the nature of his or her diagnosis, understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form.

Exclusion Criteria:

* Previous history of head and neck cancer.
* Prior acupuncture within the past month.
* Pre-existing active oral infection
* Life expectancy is < 3 months.
* Plan to go on experimental drug for head and neck cancer in the next 14 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ting Bao, MD, DABMA, Principal Investigator — University of Maryland Marlene & Stewart Greenebaum Cancer Center
Locations (1):
- University of Maryland Marlene & Stewart Greenebaum Cancer Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: University Medical Centers and Hospital Based Oncology Programs recruited participants from January 2013 until June 2014.
Pre-assignment Details: Four participants were enrolled, with three randomized to receive acupuncture and one randomized to receive standard medical care.
Period: Overall Study
Arm/Group | Acupuncture With Seirin® Needles | Usual Medical Care
Started | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture With Seirin® Needles | Usual Medical Care | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Customized [Median (Full Range); unit: years] | 63 [53 to 73] | 55 [55 to 55] | 63 [53 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Side Effects of Acupuncture Treatment
Description: All acupuncture side effects will be recorded
Time Frame: 16 weeks
Population: Zero participants analyzed due to early termination of study.
Arm/Group | Acupuncture With Seirin® Needles | Usual Medical Care
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Patients Completing Acupuncture Treatment
Description: Feasibility is defined as greater than 80% patients in the trial completing at least 4 acupuncture sessions.
Time Frame: 16 weeks
Population: Zero participants analyzed due to early termination of study.
Arm/Group | Acupuncture With Seirin® Needles | Usual Medical Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Acupuncture With Seirin® Needles | Usual Medical Care
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/1

LIMITATIONS AND CAVEATS:
The PI left the institution before the end of the study; therefore the study was withdrawn in clinicaltrials.gov and IRB closed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes